CLINICAL TRIAL: NCT02410187
Title: Stereotactic Body Radiotherapy for Extra-cranial Oligorecurrent Tumor: Randomized Phase II Clinical Trial
Brief Title: SBRT for Extra-cranial Oligorecurrent Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Mi-Sook Kim, Staff of Dept. of Radiation Oncology, Korea Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-1503-001-002
Record Dates: First submitted 2015-03-20; First posted 2015-04-07 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Recurrent Cancer
Keywords: stereotactic body radiotherapy
MeSH Terms: conditions — Recurrence | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): systemic therapy+palliative RT
  Interventions: Drug: systemic therapy (chemotherapy, hormon therapy, target therapy etc); Radiation: palliative RT
- Arm 2 (Experimental): systemic therapy+SBRT
  Interventions: Radiation: SBRT; Drug: systemic therapy (chemotherapy, hormon therapy, target therapy etc)

INTERVENTIONS:
Radiation: SBRT — 10 Gy x 3 - 20 Gy x 3 (BED 60Gy-180 Gy) or 8 Gy x 4 - 17 Gy x 4 (BED 58-184 Gy)
  Other Names: VMAT (Volumetric Modulated Arc Therapy )
  Arms: Arm 2
Drug: systemic therapy (chemotherapy, hormon therapy, target therapy etc) — Physicians can choose all the options available chemotherapy, hormon therapy, target therapy etc.
  Use of chemotherapy schemes containing potent enhancers of radiation damage (e.g. gemcitabine,adriamycin) are discouraged within the first month after SBRT.
  Other Names: chemotherapy, hormon therapy, target therapy etc.
Radiation: palliative RT — fraction size of RT = < 3 Gy
  Other Names: conventional fractionation RT
  Arms: Arm 1

SUMMARY:
Clinical experience has shown that metastasis can often be limited in number and location, and thus amenable to local treatment. The term oligometastasis describes an intermediate state of cancer spread between localized disease and widespread metastasis. The implication of such an intermediate state is that the disease can be cured by using metastasis-directed therapy. Historically, in some patients with oligometastases in the liver or lungs, surgical resection was often indicated, as abundant evidence suggested it could improve progression-free or overall survival. Recently, several studies have reported promising outcomes of >80% local control with Stereotactic Body Radiotherapy (SBRT) in patients with lung or liver oligometastases. Nonetheless, very few studies have focused on non-liver, non-lung extracranial oligometastatic lesions treated with SBRT, and such studies have limitations of a retrospective nature and small sample sizes.Because allmost studies are based on single-arm studies without appropriate controls, the level of evidence to support SBRT is weak. Randomized trials are therefore necessary to establish the utility of SBRT for oligometastatic disease.

This study is designed as a randomized phase II study. Patients will be randomized between current standard treatment (Arm 1) versus standard treatment +SBRT (Arm 2) to all known disease.

ELIGIBILITY:
Inclusion Criteria:

* age <18 years old
* ECOG score: 0-2
* number of distant metastases: 1-5
* all cancers (except lymphoma, myeloma, and germ cell tumor)
* status of primary lesion: cured
* pathologically confirmed cancer
* life expectancy: over 6 months

Exclusion Criteria:

* recurrent lesion which had been treated by radiotherapy
* complete response after systemic therapy
* patients who cannot be treated with SBRT due to any reason.
* pregnancy or breast-feeding
* malignant pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
disease progression free survival rate | 2 years

SECONDARY OUTCOMES:
overall survival rate | 2 years
local control rate | 2 years
Number of participants with radiation induced acute or late toxicity | 2 years
  Acute and late toxicities would be evaluated using the Common Terminology Criteria of Adverse Events (CTCAE) version 4.0 and the Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer (RTOG/EORTC) radiation morbidity criteria, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Sook Kim, M.D. Ph.D., Study Chair — mskim@kirams.re.kr